CLINICAL TRIAL: NCT03220633
Title: A Double-Blind, Placebo-Controlled, Phase I Study To Assess Safety, Tolerability And Pharmacokinetics Of Single/Multiple Ascending Doses Of ATB-346 Orally Administrated In Healthy Male And Female Subjects
Brief Title: Study To Assess Safety, Tolerability And PK Of ATB-346 In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Antibe Therapeutics Inc. (Industry)
Collaborators: Algorithme Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATB-346-101
Record Dates: First submitted 2015-01-06; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — 2-(6-methoxy-napthalen-2-yl)-propionic acid 4-thiocarbamoyl-phenyl ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ATB-346 (Experimental): Subjects given single dose (SAD cohorts) or multiple doses over a 14 day period (MAD cohorts) of ATB-346.
  Interventions: Drug: ATB-346
- Placebo (Placebo Comparator): Subjects given single dose (SAD cohorts) or multiple doses over a 14 day period (MAD cohorts) of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATB-346
  Arms: ATB-346
Drug: Placebo
  Arms: Placebo

SUMMARY:
A double-blind, placebo-controlled, phase I study to assess safety, tolerability and pharmacokinetics of single/multiple ascending doses of atb-346 orally administered in healthy male and female subjects.

DETAILED DESCRIPTION:
Single ascending doses of ATB-346 given to multiple cohorts followed by multiple ascending doses of ATB-346 given to multiple cohorts in order to assess its safety, tolerability, and pharmacokinetics. A single dose cohort was also conducted to assess the effect of food on the drug's characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Availability for the entire study period
2. Motivated volunteer and absence of intellectual problems likely to limit the validity of consent to participate in the study or the compliance with protocol requirements; ability to cooperate adequately; ability to understand and observe the instructions of the physician or designee
3. Healthy male or female subjects aged between 18 and 55 years, inclusive, at the time of informed consent
4. Body mass index (BMI) greater than or equal to 18.50 kg/m2 and below 30.00 kg/m2
5. Non- or ex-smokers. An ex-smoker is defined as someone who completely stopped smoking for at least six months before Day 1 of this study
6. Clinical laboratory values within the laboratory's stated normal range; if not within this range, these must be without any clinical significance
7. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on physical examination and/or clinical laboratory evaluations (hematology, general biochemistry, electrocardiogram [ECG], and urinalysis)
8. Willingness to adhere to the protocol requirements as evidenced by the informed consent form (ICF) duly read, signed and dated by the volunteer
9. A female volunteer must meet one of the following criteria:

   * If of childbearing potential - agrees to use one of the accepted contraceptive regimens from at least 28 days prior to the first drug administration, during the study and for at least 60 days after the last dose. An acceptable method of contraception includes one of the following:

     * Abstinence from heterosexual intercourse
     * Systemic contraceptives (birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch)
     * Intrauterine device (with or without hormones)
     * Condom with spermicide
   * If of non-childbearing potential - should be surgically sterile (i.e. has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or in a menopausal state (at least one year without menses)
10. A male volunteer with sexual partners who are pregnant, possibly pregnant, or who could become pregnant must meet the following criterion:

    * Participant is inapt to procreate, defined as surgically sterile (i.e. has undergone a vasectomy, it must be at least 6 months since the surgery)
    * Participant agrees to use of the accepted contraceptive regimens from first drug administration until 3 months after the last drug administration. An acceptable method of contraception includes one of the following:

      * Abstinence from heterosexual intercourse.
      * Condom with spermicide.

Exclusion Criteria:

1. Females who are pregnant or breastfeeding
2. Seated pulse rate less than 50 Beats per Minute (bpm) or more than 100 bpm at screening
3. Seated blood pressure below 100/60 mmHg or higher than 140/90 mmHg at screening
4. History of significant hypersensitivity to naproxen, other non-steroidal anti-inflammatory agents, or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
5. Presence of significant gastrointestinal, liver, or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs or know to potentiate or predispose to undesired effects
6. Presence of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic, or dermatologic disease
7. Suicidal tendency, history of/or disposition to seizures, state of confusion, clinically relevant psychiatric diseases
8. Presence of out-of-range cardiac interval (PR < 110 msec, PR > 200 msec, QRS < 60 msec, QRS >110 msec and QTc > 440 msec) on the screening ECG or other clinically significant ECG abnormalities
9. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (>3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
10. Any clinically significant illness in the previous 28 days before Day 1 of this study
11. Use of any enzyme-modifying drugs, including strong inhibitors of CYP enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem, and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin and St John's Wort) in the previous 28 days before Day 1 of this study
12. Any history of tuberculosis and/or prophylaxis for tuberculosis
13. Positive urine screening of alcohol and/or drugs of abuse
14. Positive results to HIV Ag/Ab Combo, Hepatitis B surface Antigen (HBsAg) or anti-Hepatitis C Virus (HCV) tests
15. Females who are pregnant according to a positive serum pregnancy test
16. Volunteers who took an Investigational Product (in another clinical trial) in the previous 28 days before Day 1 of this study or who have already participated in this clinical study
17. Volunteers who donated 50 mL or more of blood in the previous 28 days before Day 1 of this study
18. Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc) in the previous 56 days before Day 1 of this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Within one week following single dose administration or within one week following the final dose after two weeks of treatment regimen
  Serum chemistry and hematology laboratory measures

CONTACTS AND LOCATIONS:
Locations (1):
- Algorithme Pharma, Montreal, Quebec, Canada